CLINICAL TRIAL: NCT00338624
Title: A Double-Blind, Randomized, Parallel Group Trial of Ditropan XL (Oxybutynin Chloride) Extended Release Tablets or Placebo in Combination With FLOMAX (Tamsulosin Hydrochloride) for the Treatment of Lower Urinary Tract Symptoms.
Brief Title: An Effectiveness and Safety Study Comparing Oxybutynin Chloride Plus FLOMAX (Tamsulosin HCl) and Placebo Plus FLOMAX (Tamsulosin HCl) for the Treatment of Lower Urinary Tract Symptoms.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004675
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2010-04

CONDITIONS: Urination Disorders
Keywords: lower urinary tract symptoms; DITROPAN XL; oxybutynin extended release tablets
MeSH Terms: conditions — Urination Disorders; Lower Urinary Tract Symptoms

INTERVENTIONS:
Drug: oxybutynin chloride extended release

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of oxybutynin extended release tablets 10 mg plus tamsulosin HCl 0.4 mg in the treatment of lower urinary tract symptoms as measured by change of the total International Prostate Symptom Score (I-PSS) from baseline to Week 12 or the Final Visit.

DETAILED DESCRIPTION:
The objective of this double-blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage), randomized (patients are assigned different treatments based on chance), parallel group trial is to evaluate the safety and effectiveness of oxybutynin extended release tablets 10 mg per day for 12 weeks in conjunction with an alpha-blocker for the treatment of lower urinary tract symptoms (LUTS). The hypothesis of the study is that oxybutynin extended release tablets 10 mg plus tamsulosin 0.4 mg will be more effective than tamsulosin 0.4 mg plus placebo in the treatment of lower urinary tract symptoms as measured by change of the total International Prostate Symptom Score (I-PSS) from baseline to Week 12 or the Final Visit. Safety assessments include Peak Flow Rate (PFR) and Post-Void Residual (PVR) volume, adverse events, vital signs and physical exams. Patients will receive oxybutynin extended release 10 mg plus tamsulosin 0.4 mg or placebo plus tamsulosin 0.4 mg every day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lower urinary tract symptoms with urgency and frequency with or without urge incontinence
* have had at least 4 weeks of 0.4 mg/day tamsulosin therapy
* an International Prostate Symptom Score (I-PSS) >=13
* irritative component I-PSS score >= 8
* max flow >= 8ml/sec with voided volume >= 125 ml, post-void residual volume <= 150 ml on two occasions.

Exclusion Criteria:

* Clinically significant medical problems or other organ abnormality or pathology
* Prostate-Specific Antigen (PSA) >= 4 ng/ml
* history of inability to empty bladder completely or not at all
* uncontrolled narrow angle glaucoma
* history of any prostate surgery or treatment
* history of significant gastrointestinal problems.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2004-05; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change of the total International Prostate Symptom Score (I-PSS) from baseline to Week 12 or the Final Visit.

SECONDARY OUTCOMES:
At all timepoints assessed and final visit: I-PSS (total score, irritative component score, quality of life score); Symptom Problem Index score; Urgency and frequency scales scores; Incontinence Indicator scale score

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- See also: An effectiveness and safety study comparing oxybutnin chloride plus FLOMAX (tamsulosin HCL) and placebo plus FLOMAX (tamsulosin HCL) for the treatment of lower urinary tract symptoms — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1088&filename=CR004675_CSR.pdf